CLINICAL TRIAL: NCT05900492
Title: Incidence of Uterine Cesarean Scar Niche After Cesarean Delivery and Assessment of Its Risk Factors
Brief Title: Incidence of Uterine Cesarean Scar Niche After Cesarean Delivery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Abdallah Mohamed Salem, principle investigator/Lecturer of Gynecology and obstetrics Faculty of medicine Beni-Suef University, Beni-Suef University
Other Study IDs: cesarean scar niche R.F
Record Dates: First submitted 2023-06-04; First posted 2023-06-12 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Cesarean Section; Dehiscence
MeSH Terms: interventions — Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- previous 1 cesarean section: patient who had her first Cesarean section
  Interventions: Procedure: cesarean section
- previous 2 cesarean sections: patient who had her second Cesarean sections
  Interventions: Procedure: cesarean section
- previous 3 or more cesarean sections: patient who had 3 or more Cesarean sections
  Interventions: Procedure: cesarean section

INTERVENTIONS:
Procedure: cesarean section — caesarean delivery, is the surgical procedure by which one or more babies are delivered through an incision in the mother's abdomen

SUMMARY:
To assess the incidence of cesarean scar niche and its risk factors in a prospectively collected population.

DETAILED DESCRIPTION:
It will be carried out in Gynecology and Obstetrics department in Beni-Suef University Hospital using Ultrasound:

Six months after the cesarean delivery, participants will be invited to the gynecologic outpatient clinic or department for ultrasound (US) examination to detect the presence of the niche.

Women without contraception will be examined during the follicular phase of the menstrual cycle to avoid an eventual early pregnancy. Otherwise, a random phase of the menstrual cycle will be accepted. Women who are pregnant at the time of US will be excluded. Women will be examined in the lithotomy position with an empty bladder. The uterus will be examined in a standardized way, with trans-vaginal US performed first.

For the diagnosis of cesarean scar niche (defined as an anechoic defect in the anterior wall of the lower uterine segment, communicating with the endometrial cavity),we will use a predetermined definition of a defect at least 2.0 mm deep

ELIGIBILITY:
Inclusion Criteria:

1. Delivery by cesarean section.
2. More than 6 months after delivery.
3. Cesarean section by senior resident or assistant lecturer.

Exclusion Criteria:

1. Single layer technique in uterine closure.
2. Uterine anomaly.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will include women recruited from the outpatient obstetrics clinic or emergency room after proper counseling.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
the incidence of cesarean scar niche among cesarean deliveries | 6 months after delivery
  number of cases develop cesarean scar niche after cesarean deliveries

SECONDARY OUTCOMES:
risk factors that affect the development of the niche. | within 1 month of delivery
  age- BMI- post operative infection - PROM(preterm rupture of membrane)

CONTACTS AND LOCATIONS:
Overall Officials: sara M salem, MD, Principal Investigator — Faculty of Medicine Beni-Suef University
Locations (1):
- Beni-suef university Hospital, Banī Suwayf, Beni Suweif Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided